CLINICAL TRIAL: NCT06366607
Title: Medication Safety Climate: Managing High-alert Medication Administration and Errors Among Nurses in Intensive and Critical Care Units
Brief Title: Managing High-alert Medication Administration and Errors
Status: Completed | Type: Observational
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Nagah Abd El-Fattah Mohamed Aly, Assistant professor of Nursing administration, Matrouh University
Other Study IDs: 0306066
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Knowledge; Practice Nurse's Scope; Competence; Nurse's Role; Error Disclosure
Keywords: Medication safety climate; Managing, High-alert medication; Administration; Errors; Nurses' role

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nurses: Nurses worked in surgical intensive and critical care units
  Interventions: Other: high-alert medication administration

INTERVENTIONS:
Other: high-alert medication administration — high-alert medication administration

SUMMARY:
High-alert medications are drugs that may lead to serious harm when they are wrongly administered to patients. Safe medication administration is the crucial role of nursing staff.

DETAILED DESCRIPTION:
High-alert medications are drugs that may lead to serious harm when they are wrongly administered to patients. Safe medication administration is the crucial role of nursing staff. This study aims to investigate the relationships between medication safety climate and nurses' knowledge about high-alert medications with managing their administration and errors.

ELIGIBILITY:
Inclusion Criteria:

* Nurses

  * willing to participate in the study
  * work in surgical intensive and critical care units
  * Sign a consent

Exclusion Criteria:

- Nurses

* Work in outpatient units and other units
* Did not sign a consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A sample of 300 nurses was enrolled in the current study. The nurses were willing to participate in the study and provided their agreement by informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure nurses' knowledge about high-alert medication administration | one month
  Nurses' knowledge about high-alert medication administration as assessed binary scale.
Questionnaire to measure medication safety climate | one month
  Medication safety climate as assessed using five-point Likert scale ranging from strongly disagree (1 point) to strongly agree (5 points).
Questionnaire to measure nurses' competency | one month
  Nurses' competency during the administration of high-alert medications as assessed using five- Likert scales ((0 = not appropriate at all in administering high-alert medications up to 4 = very often appropriate in administering high-alert medications)
observational check list to measure nurses' practice during administration of high-alert medications | one month
  Observing nurses' practice during the administration of high alert medications as assessed using five Likert scales (0=inappropriate practice up to 4=appropriate practice)
Questionnaire to measure errors associated with administering high-alert medications | one month
  Errors associated with administering high-alert medications as assessed using a binary scale ( Yes=1 , No=0)

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abd El-Fattah Mohamed Aly, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University, Egypt; Wael M. Lotfy, Ph.D, Study Director — Faculty of Nursing, Matrouh University, Egypt; Safaa M. El-Shanawany, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Maha Ghanem, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Hanaa Abbass, Ph.D, Principal Investigator — Psychatric Nursing and Mental health , Faculty of Nursing, Alexandria University, Egypt; Maysa Elbiaa, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University , Egypt
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No